CLINICAL TRIAL: NCT04284878
Title: Lymphoid Tyrosine Phosphatase Gene Polymorphisms in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Refaat Ali, doctor, Assiut University
Other Study IDs: LYP polymorphisms in IBD
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — gene polymorphisms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: patients with inflammatory bowel disease
  Interventions: Genetic: PCR-RFLP
- B: healthy subjects
  Interventions: Genetic: PCR-RFLP

INTERVENTIONS:
Genetic: PCR-RFLP — PCR-Restriction fragment length polymorphism

SUMMARY:
This study aims:

1. To investigate the association between single nucleotide polymorphisms of PTPN22 gene (rs2476601, rs33996649 and rs2488457) and inflammatory bowel disease.
2. To correlate the relation between the studied SNPs and disease activity /response to therapy.

DETAILED DESCRIPTION:
The inflammatory bowel diseases (IBD) are chronic inflammatory disorders of the gastrointestinal tract that manifests as Crohn's disease (CD) and Ulcerative colitis (UC), clinically characterized by periods of remission interrupted by episodes of clinical disease activity (Zallot et al., 2013). Patients with IBD display some common symptoms such as severe diarrhea, pain, fatigue and weight loss , but the localization is slightly different: whereas CD affects the whole gastrointestinal tract, UC primarily affects the distal intestine and ileum (De Lange et al., 2015).

Lennard-Jones et al. have defined macroscopic and microscopic criteria to establish the diagnosis of Crohn's disease. The macroscopic diagnostic tools include physical examination, endoscopy and radiology. Microscopic features can be assessed on mucosal biopsy and/or operative specimen. The diagnosis depends on the finding of discontinuous and often granulomatous intestinal inflammation (Lennard-Jones et al., 1997). Diagnosis of ulcerative colitis is based on history, endoscopic appearances, histopathology of multiple mucosal biopsies and appropriate radiology (Silverberg et al., 2005, Satsangi et al., 2006).

The incidence pattern of UC has changed over the last two decades, with incidence continuing to rise in the West and rising incidence in previously low incidence areas such as Asia and the Middle East (0.15- 6.5 per 100,000)(Ng et al., 2017). Marked increase in UC diagnoses was noted over a 15-year period (1995-2009). In Cairo University, 17 cases were recorded in 1995-1999 and 76 cases were recorded in 2005-2009 (Esmat et al., 2014).

Both CD and UC are complex diseases genetically, in which hundreds of independent genetic loci contribute to disease susceptibility (Norouzinia et al., 2015) . Nevertheless, the molecular mechanisms and functions of many IBD associated genes remain unknown. In addition to genetics, IBDs are powerfully influenced by microbiological and environmental aspect (Norouzinia et al., 2017).

Genome-wide association studies (GWAS) have allowed a better understanding of IBD thus, several genetic susceptibility loci have been identified for UC and CD (Yamamoto-Furusho et al., 2015). Among the genetic factors involved, there are several polymorphisms in molecules of the Immune system associated with either susceptibility or protective effects to IBD progression, but even with contradictory associations, mainly depending on the onset (adult or pediatric), sample size differences and on the ethnicity-dependent genetic background (Neuman et al., 2012, Ng et al., 2012, Peng et al., 2017, Girardelli et al., 2018).

PTPN22 protein contains three domains, including: an N-terminal PTP catalytic domain; an interdomain region; and a C-terminal domain with four proline-rich regions that function as motifs for interaction with other protein (Stanford et al., 2014).Tyrosine phosphatase is involved in maintaining intestinal epithelial barrier function, regulating autophagosome function and immune responses to invading bacteria in intestinal cells, limiting pro-inflammatory cytokine secretion in the intestine as well as controlling differentiation and function of CD4+ T-cells in vivo (Spalinger et al., 2015). The lymphoid tyrosine phosphatase (Lyp) encoded by PTPN22 plays a critical role as a negative regulator of T-cell activation by dephosphorylating T-cell receptor activation dependent kinases (Csk kinase) (Cloutier et al., 1999). PTPN22 is a critical regulator of the (Nod Like Receptor Family Pyrine Domain Containing 3 ) NLRP3 inflammasome by controlling NLRP3 tyrosine phosphorylation . Further, PTPN22 controls NLRP3-mediated IL-1beta secretion in an autophagy dependent manner (Yilmaz et al., 2018) .

PTPN22 gene is located on the short arm of Chromosome 1 (1p13.2). There are 24 exons in the gene (NCBI website).About 21 SNPs were found in PTPN22 gene (rs1310182, rs3789604, rs33996649, rs1217414, rs2476601, rs12760457, rs2488457,,,,etc).SNP rs2476601 (C1858>T) in exon 14 results in the substitution of arginine 620 with a tryptophan residue in the protein product (referred to as 620W variant) (Spalinger et al., 2016). SNP rs33996649 (G788>A) in exon 10 mediates substitution of arginine 263 with a glutamine residue (referred to as 263Q variant) and affects the ability of Lyp to interact with the Csk kinase, thus avoiding the formation of the complex and the resulting suppression of T-cell activation(Hedjoudje et al., 2017) . SNP rs2488457 (G -1123>C) is located in the promoter region (Chen et al., 2013).A transcription factor binding site for activator protein 4 (AP-4) at position -1123 is predicted in the presence of the G allele rather than the C allele (Jüliger et al., 2003).

Contradictory results have been published regarding the association of PTPN22 gene SNPs with IBD (Bank et al., 2014, Sfar et al., 2010, Chen et al., 2013, Latiano et al., 2007, Diaz-Gallo et al., 2011, Wagenleiter et al., 2005, Zaid et al., 2018, Sadr et al., 2019).

In Egypt studies were done regarding the association of PTPN22 gene SNPs with{ Type1 DM (El-Kafoury et al., 2014), ITP (Anis et al., 2011) ,SLE (Elghzaly et al., 2015) , Alopecia Areata (El-Zawahry et al., 2013) and RA (Salama et al., 2014) }.

Uptodate , no studies were published regarding the association of PTPN22 gene SNPs with IBD in egyptians.

ELIGIBILITY:
Inclusion Criteria:

* patients with inflammatory bowel disease

Exclusion Criteria:

* Patients with systemic autoimmune diseases (RA,SLE) will be excluded from the study .

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: IBD Patients will Diagnosed according to established guidelines for UC/CD . Phenotype characteristics of UC and CD were defined according to the Montreal classification . The clinical disease activity will be assessed using the Montreal classification of UC disease activity and Crohn's Disease Activity Index (CDAI) for CD
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Association between single nucleotide polymorphisms of Lymphoid Tyrosine Phosphatase gene (rs2476601, rs33996649 and rs2488457) and inflammatory bowel disease | baseline
  Three single nucleotide polymorphisms in the lymphoid tyrosine phosphatase gene(SNP (G788>A) in exon10, SNP (C1858>T) in exon 14 and SNP (G -1123>C) in the promoter region ) will be assessed in 100 patients diagnosed as inflammatory bowel disease and 100 healthy subjects by Polymerase Chain Reaction-Restriction Fragment Length Polymorphism (PCR-RFLP) to detect association between these polymorphisms and inflammatory bowel disease

SECONDARY OUTCOMES:
To correlate the relation between the studied SNPs and disease activity /response to therapy. | baseline
  Serum Erythrocyte Sedimentation Rate ,C-Reactive Protien ,Anti Nuclear Antibody ,Antineutrophil Cytoplasmic Antibody (ANCA) and Anti Saccharomyces Cerevisiae (ASCA) and fecal calprotectin will be done to all patients.The three investigated polymorphisms in LYP will be correlated with the markers of disease activity and IBD patients response to therapy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norouzinia M, Chaleshi V, Alizadeh AHM, Zali MR. Biomarkers in inflammatory bowel diseases: insight into diagnosis, prognosis and treatment. Gastroenterol Hepatol Bed Bench. 2017 Summer;10(3):155-167. PMID 29118930